CLINICAL TRIAL: NCT00255528
Title: Dose Ranging, Safety and Tolerability of TOPROL-XL® (Metoprolol Succinate) Extended-Release Tablets (Metoprolol CR/XL) in Hypertensive Pediatric Subjects: A Multicenter, Double-Blind, Placebo-Controlled, Randomized, Parallel-Group Study
Brief Title: Dose Ranging, Safety and Tolerability of TOPROL-XL® Extended-Release Tablets in Hypertensive Pediatric Subjects
Acronym: 307A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D4020C00033; 307A; SH-MET-0033
Record Dates: First submitted 2005-11-17; First posted 2005-11-21 (Estimated); Last update posted 2007-03-20 (Estimated); Status verified 2007-03

CONDITIONS: Hypertension
Keywords: Pediatric hypertension
MeSH Terms: conditions — Hypertension | interventions — Metoprolol

INTERVENTIONS:
Drug: metoprolol succinate

SUMMARY:
This was a 4-week, multicenter, double-blind, placebo-controlled, randomized, parallel-group study to determine the antihypertensive dose range, efficacy, safety and tolerability of TOPROL-XL ® (metoprolol succinate) extended-release tablets (metoprolol CR/XL) in hypertensive pediatric subjects. The study population included school age children (age 6 to < Tanner Stage 3) and adolescents (> Tanner Stage 3 to age 16) of both genders. No more than 50% of the randomized subjects could be adolescents (> Tanner Stage 3 to 16 years old). Since response to some therapies in adult hypertension appears to be different in black and non-black populations, recruitment was aimed at a mixture of black and non-black children. The design included a 1-week screening period (for treatment naive subjects), a 1-week single-blind placebo run-in period, and a 4-week double-blind treatment period. Eligible subjects were randomized to the double-blind period with a once daily oral dose of metoprolol CR/XL to one of three target doses: 0.2, 1.0 and 2.0 mg/kg, or placebo. Dosing was weight adjusted. The dose range for this study was 12.5 to 200 mg daily. Subjects were closely monitored and evaluated at the end of Weeks 1, 2, 3 and 4 during the double-blind treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 6 and 16 years inclusive at the time of screening.
* Have a negative urine pregnancy test, if female of childbearing potential.
* Have a signed informed consent by a parent or a legal guardian and an assent form signed by the subject (if applicable).
* Have hypertension that is either:

  1. Newly diagnosed and untreated with a mean sitting SBP or DBP above the 95 th percentile on three consecutive office visits, or
  2. Previously diagnosed and currently treated with antihypertensive therapy at Visit 1, then at Visit 3 (off treatment) have a mean sitting SBP or DBP above the 95 th percentile.
* Have the ability to swallow tablets.

Exclusion Criteria:

* Have secondary hypertension due to coarctation of aorta, pheochromocytoma, hyperthyroidism or Cushing's syndrome.
* Have SBP or DBP greater than 20 (SBP) or 10 (DBP) mm Hg above the 95th percentile using height adjusted charts for age and gender.
* Have a heart rate < 55 beats per minute at randomization.
* Have a history of asthma and/or recurring pulmonary disease or infections.
* Have a history of cystic fibrosis.
* Have a known hypersensitivity reaction to beta-blockers.
* Have a known bleeding, coagulation or platelet disorder that can interfere with blood sampling.
* Have a history of Insulin Dependent Diabetes Mellitus.
* Be in any situation or have any condition which, in the opinion of the investigator or sponsor, may interfere with participation in the study or produce a significant risk to the subject or interfere with the assessment of safety and efficacy endpoints.
* Have received any investigational agent for any therapeutic reason within 30 days prior to receiving study medication.
* Have a clinically significant cardiac valvular disease.
* Have a diagnosis of heart failure.
* Have clinically significant arrhythmia. This is defined as any arrhythmia requiring medical therapy or that causes symptoms.
* Atrioventricular (AV) conduction disturbance, ie, second or third degree AV block.
* Be unable or unwilling to comply with the study requirements.
* Be non-compliant during the single-blind placebo run-in period of the study as defined by missing three or more doses between study visits.
* Have impaired liver function defined as either acute liver disease or chronic liver disease with persistent liver enzyme values greater than one and one half times the upper limit of the normal range for AST or ALT.
* Have a known history of bilateral renal artery stenosis, or unilateral renal artery stenosis to a single kidney. Nephrotic subjects who are not in remission should be excluded.
* Be pregnant or breast-feeding an infant.
* Currently taking medications known to inhibit CYP2D6, such as quinidine, fluoxetine, paroxetine and propafenone.
* Currently taking catecholamine-depleting medications such as reserpine. For any subject who is currently taking medications known to inhibit CYP2D6 or any catecholamine-depleting medication, the sponsor must be contacted to assess feasibility for inclusion into the study.
* Currently taking any selective serotonin re-uptake inhibitors (SSRIs) or atypical antipsychotic medication.
* Have a history of alcohol or drug abuse, or have a positive urine screen for drugs of abuse or alcohol.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 144
Dates: Start 2002-07

PRIMARY OUTCOMES:
To evaluate the dose range, safety, and tolerability of metoprolol CR/XL in hypertensive pediatric subjects, based on the change in sitting SBP from baseline to the end of treatment.

SECONDARY OUTCOMES:
Slope of placebo-corrected changes in sitting DBP: baseline to end of treatment as a function of target dose. Differences in mean change: baseline to end of treatment comparing each active group to placebo for sitting SBP and DBP.
Safety profile

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Toprol Medical Science Director, MD, Study Director — AstraZeneca
Locations (31):
- United States (30):
  - Research Site, Little Rock, Arkansas
  - Research Site, Bellflower, California
  - Research Site, Beverly Hills, California
  - Research Site, Los Angeles, California
  - Research Site, Orange, California
  - Research Site, Hartford, Connecticut
  - Research Site, Wilmington, Delaware
  - Research Site, Gainsville, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Tampa, Florida
  - Research Site, Honolulu, Hawaii
  - Research Site, Chicago, Illinois
  - Research Site, Louisville, Kentucky
  - Research Site, Livingston, New Jersey
  - Research Site, New Hyde Park, New York
  - Research Site, The Bronx, New York
  - Research Site, Durham, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Landsdale, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Greenville, South Carolina
  - Research Site, Beaumont, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Norfolk, Virginia
- Research Site, Santo Domingo, Dominican Republic

REFERENCES:
- [Derived] Batisky DL, Sorof JM, Sugg J, Llewellyn M, Klibaner M, Hainer JW, Portman RJ, Falkner B; Toprol-XL Pediatric Hypertension Investigators. Efficacy and safety of extended release metoprolol succinate in hypertensive children 6 to 16 years of age: a clinical trial experience. J Pediatr. 2007 Feb;150(2):134-9, 139.e1. doi: 10.1016/j.jpeds.2006.09.034. PMID 17236889